CLINICAL TRIAL: NCT04629430
Title: Effects of Prebiotics on Gut Microbiome in Patients Undergoing Stem Cell Transplants
Brief Title: Effects of Prebiotics on Gut Microbiome in Patients Undergoing HSCT
Acronym: HCTDiet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Indumathy Varadarajan, MD, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR 200296
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Multiple Myeloma; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Non Hodgkin Lymphoma; Acute Lymphocytic Leukemia; Hodgkin Lymphoma; Hodgkin Disease; Myelofibrosis; Myelodysplastic Syndromes; Myeloproliferative Neoplasm; Sickle Cell Disease; Mantle Cell Lymphoma
Keywords: hematopoietic stem cell transplant; stem cell transplant; bone marrow transplant; GI microbiome
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Primary Myelofibrosis; Myelodysplastic Syndromes; Myeloproliferative Disorders; Anemia, Sickle Cell; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prebiotic diet (Experimental): 2 servings a day of pre-biotics every day from start of conditioning regimen for HSCT through 100 days following HSCT
  Interventions: Other: Pre-biotic foods/drinks

INTERVENTIONS:
Other: Pre-biotic foods/drinks — 2 servings per day

SUMMARY:
The purpose of this study is to see whether hematopoietic stem cell transplant (HSCT) patients can consistently eat a diet rich in prebiotics. This type of diet may be helpful in maintaining diversity in the gastrointestinal (GI) system and therefore potentially decreasing risk of other GI problems.

DETAILED DESCRIPTION:
Maintaining gastrointestinal (GI) microbiome diversity has been shown to improve treatment related mortality in HSCT patients. Interventions to improve GI microbial diversity could be beneficial to this patient population. Diets rich in prebiotics have been shown to increase gut microbial diversity and improve symptoms in other gastrointestinal diseases. Prebiotics are non-digestible carbohydrates that promote growth of commensal organisms in the gut by providing nutrition. Some examples are brown rice, green apples, and tomatoes. Our theory is that consuming a diet rich in prebiotics pre- and during the first 100 days following HSCT will help to reduce acute graft versus host disease (aGVHD) overall, and specifically acute GI GVHD, and clostridium difficile (C.Diff). Participants will be encouraged to eat at least 2 servings of a prebiotic-rich food from time of admission for HSCT through 100 days following HSCT and will be clinically monitored, including for acute GVHD, acute GI GVHD and C.Diff. Stool samples will be collected from all participants about once every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Agreement to adhere to Lifestyle Considerations(prebiotic diet) throughout study duration
2. Adults (≥18 yrs of age)
3. Able to provide informed consent
4. Are willing/able to incorporate the required foods in their diet
5. Eligible, suitable and planning to undergo a stem cell transplant:

   1. Either allogeneic or autologous
   2. With any conditioning regimen (e.g. both myeloablative and reduced intensity conditioning)
   3. Matched related, matched unrelated, haplo-identical and cord blood transplants will be included.

Exclusion Criteria:

1. Patients undergoing a second allogeneic or autologous transplant or an allogeneic transplant after an autologous transplant.
2. Anticipation of requirement of broad spectrum antibiotics 1 week prior to admission for HSCT (through HSCT)
3. Patients with any prior history of C.Diff infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Frequency of participants ingesting the required diet | From initiation of conditioning regimen for HSCT through 100 days following HSCT
  Frequency of participants reporting ingesting at least 2 servings of prebiotics on ≥ 80% of study days

SECONDARY OUTCOMES:
Incidence and severity of acute GVHD (aGVHD) and acute GI GVHD | Within the first 100 days following HSCT
  Stage and grade of aGVHD (allogeneic HSCT participants only)
Incidence of CDiff infection | Within the first 100 days following HSCT
  Number of people diagnosed with CDiff during the time frame
Patient weight | From initiation of conditioning regimen for HSCT through 100 days following HSCT
Number of days to neutrophil engraftment | From initiation of conditioning regimen for HSCT through 100 days following HSCT
  Absolute neutrophil count >1000 for 1 day or > 500 for 3 consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: Indumathy Varadarajan, Principal Investigator — Assistant Professor
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No